CLINICAL TRIAL: NCT05548816
Title: Prevalence of Subacromial Impingement Among Egyptian Swimmers a Cross Sectional Survey Study.
Brief Title: Prevalence of Subacromial Impingement Among Egyptian Swimmers
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Morog Galal Nadim, Principal investigator, Cairo University
Other Study IDs: 15121993
Record Dates: First submitted 2022-07-12; First posted 2022-09-21 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Swimmers; Swimmer's shoulder; Subacromial impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Subgroup (1) Male: Includes swimmers from 12 to less than 14 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (2) Male: Includes swimmers from 14 to less than 16 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (3): Male: Includes swimmers 16 to less than 18 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (4) Male: Includes swimmers from 18 to less than 20 years
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (5) Male: (1st Team) includes swimmers from 20 - 25 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (1) Female: Includes swimmers from 12 to less than 14 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (2) Female: Includes swimmers from 14 to less than 16 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (3) Female: Includes swimmers 16 to less than 18 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (4) Female: Includes swimmers from 18 to less than 20 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .
- Subgroup (5) Female: (1st Team) includes swimmers from 20 - 25 years.
  Interventions: Other: Handheld Dynamometer , Special tests and Modified DASH questionarre .

INTERVENTIONS:
Other: Handheld Dynamometer , Special tests and Modified DASH questionarre . — A mix of tools , special tests and questionarre to help in confirming the diagnosis of subacromial impingement.
  Other Names: Special tests ( Lift-off , Neers , Hawkins and kennedy tests); Modified DASH (Disabilities of the Arm, Shoulder, and Hand) questionarre .

SUMMARY:
In the available literature, there are no prevalence studies that show the incidence of subacromial impingement in swimmers in Egypt, this should be considered as it's one of the most commonly reported injuries worldwide in swimmers. There are also no available studies to show the difference in incidence of subacromial impingement between both genders in Egypt. This study is attempting to remedy both research deficits and to reduce the literature gap and to show the prevalence rate of this injury among Egyptian swimmers in different age groups, to help prevent its widespread and to provide data for further investigations. This study would give the Egyptian swimming federation and the Ministry of youth and sports a clear idea about the prevalence rate of swimmer's shoulder at different ages in Egyptian swimmers. Most importantly, this study is to provide the physiotherapy community in Egypt data about this injury, the rate of prevalence and how to prevent it and hopefully would help in further future studies and also to apply it in different countries.

ELIGIBILITY:
Inclusion Criteria:

* 440 swimmers (males and females) , their age between 12 - 25.
* Professional swimmers only.
* Complain of anterior shoulder pain while swimming or elevation of shoulder.
* BMI will be ranged from (18.5 - 24.9 kg/m2 ).
* All swimmers are under supervision and psychologically, medically stable.
* All swimmers received a good explanation of the questionnaire and the given study.

Exclusion Criteria:

* Any swimmer who refuse to participate in the study
* Uncooperative swimmers.
* Unprofessional swimmers.
* Participants who play any other sports.
* Exclude any previous traumatic lesion.
* Exclude any form of shoulder instability.
* Take any medication that affects pain perception as NSAIDS.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Egyptian swimmers , Age ranging from 12 - 25 as mentioned in the subgroups and this study will be taken as a one shot.
  Swimmers will be collected from (Al-Ahly, Heliopolis, Shooting, El Shams, Al-zohour ,platinum , El-Nasr, Cairo ,Al-Maadi, Tala'ea Elgeish, Ittihad el shorta , El- Rowad ,Wadi-Degla, Shooting ,El Ghaba and El Geziera Sporting Clubs).
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
External / lnternal rotation ratio | 1 day
  Measured by Handheld dynamometer
Lift-off test | 1 day
  This test is performed in a standing position, with the examiner observing and testing from standing behind the patient. To perform this test, the patient is asked to place the back of the affected arm (dorsum of the hand) in the mid lumbar spine area. The testing movement involves the patient performing internal rotation (IR), by lifting the hand off the back while the examiner places pressure on the hand. The test is considered to be positive if the patient cannot resist, lift the hand off the back or if she/he compensates by extending the elbow and shoulder.
Neers test | 1 day
  Neer's sign In standing the patient's arm was passively elevated in the plane of the scapula while preventing rotation of the scapula. Reproduction of pain at the anterior edge of the acromion/lateral deltoid was considered a positive response for impingement.
Hawkins and kennedy test | 1 day
  Hawkins and Kennedy test while sitting, with the elbow flexed to 90, the patient's shoulder was passively elevated to 90 in the sagittal plane and then forcefully rotated medially. Pain indicated a positive test result.
Modified QuickDASH questionarre result | 1 day
  The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (4 items, scored 1-5) .For Example in the disability / symptoms sections , at least 10 of the 11 items must be completed for a score to be calculated.
  The assigned values for all completed responses are simply summed and averaged, producing a score out of five.This value is then transformed to a score out of 100 by subtracting one and multiplying by 25 , measures scaled on a 0-100 scale. A higher score indicates greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrilife clinic, Cairo, Egypt